CLINICAL TRIAL: NCT00035451
Title: Efficacy and Safety Evaluation of Azimilide or Sotalol vs Placebo for Treatment of Patients With Atrial Fibrillation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1999105
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — azimilide; Sotalol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): placebo tablets
  Interventions: Drug: Placebo
- 2 (Active Comparator): Sotalol
  Interventions: Drug: Sotalol
- 3 (Experimental): azimilide
  Interventions: Drug: Azimilide Dihydrochloride

INTERVENTIONS:
Drug: Azimilide Dihydrochloride — 125 mg azimilide tablets, twice a day for 6 months
  Arms: 3
Drug: Placebo — tablets, twice daily for 6 months
  Arms: 1
Drug: Sotalol — 160 mg sot twice daily for 6 months
  Arms: 2

SUMMARY:
Atrial fibrillation (abnormal rhythm in the upper chamber of the heart) is a common supraventricular arrhythmia (a type of abnormal heart rhythm) for which antiarrhythmic therapy is often prescribed. The primary goals of therapy are to maintain sinus rhythm (normal heart rhythm) and to reduce the occurrence of episodes of atrial fibrillation.

The double-blind, placebo-controlled phase of this study is designed to evaluate the efficacy and safety of oral azimilide compared with placebo and with sotalol, an antiarrhythmic drug, in maintaining sinus rhythm in patients who require cardioversion (electric shock to correct heart rhythm) to correct atrial fibrillation. Once this phase of the study is completed, a second phase with a different study design will be conducted. The second phase is an open-label, follow-up phase to the first study. The follow-up phase will continue to evaluate the long-term safety of a daily oral dose of azimilide in patients who complete the double-blind, placebo-controlled phase of this study.

ELIGIBILITY:
Inclusion criteria:

* Documented (12-lead ECG) history of symptomatic atrial fibrillation occurring between 48 hours and 6 months before screening
* Require the procedure of cardioversion (electric shock to correct abnormal rhythm)
* In the investigator's opinion, is likely to maintain sinus rhythm after cardioversion.
* Be anticoagulated according to the recommendations of the Study Group on Atrial Fibrillation of the European Society of Cardiology guidelines.

Exclusion criteria:

* Previously unsuccessful electrical cardioversions
* Failed to respond to any Class III antiarrhythmic drugs
* Qualifying arrhythmia due to acute reversible illness, acute myocardial infarction, and/or cardiac or thoracic surgery within one month prior to randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2001-02; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
To prolong the time to first symptomatic or asymptomatic AFIB, etc event | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Cuenca, MD, Study Director — Procter and Gamble
Locations (129):
- Belgium (3):
  - Clinique Generale Saint Jean Service de cardiologie, Brussels
  - Hospital Universitarie Erasme, Brussels
  - Cliniques Univeristaires UCL Mont-Godinne Avenue Theresse 1, Yvoir
- France (15):
  - Service de Cardilolgie CH du Pays d'Aix, Aix-en-Provence
  - CHR Besancon Service de cardiologie, Besançon
  - Hopital Gavriel Montpied Cardiologie-Maladie cardiovascularies, Clermont-Ferrand
  - Service de Cardiologie CHRU, Grenoble
  - Cardiologie Hopital Jean Rostand, Ivry-sur-Seine
  - Service de Cardiologie A Hopital Cardiologique, Lille
  - Service de Cardiologie Hopital Saint Philibert, Lomme
  - Cardilolgie Hopital Guillaume et Rene Laennec, Nantes
  - Service de Cardiologie Hopital Lariboisiere, Paris
  - Service de Cardiologie et Maladies Vascularies CHRU Pontchaillou, Rennes
  - Cardiologie CHRU St Etienne/Hopital Nord, Saint-Etienne
  - Centre Hospitalier General Hospital De Girac, Saint-Michel-sur-Orge
  - Cardiologie/Pavillon Baudot Centre Hospitalier Universitaire Purpan, Toulouse
  - Cardiologie A CHU Rangueil, Toulouse
  - Service de cardiologie Hopitaux de Brabois/CHRU Nancy, Vandœuvre-lès-Nancy
- Germany (24):
  - Erzgebirgskrankenhaus Klinik fur Innere Medizin, Annaberg
  - Kerckhhoff-Klinik Abteilung Klinische Pharmakologie, Bad Nauheim
  - Kardiologie Herzzentrum Osnabruck, Bad Rothenfelde
  - Dr. Schreiber Krankenhaus Neukoelin 1 Innere Rudowerstrasse, 48, Berlin
  - Franz-Volhard-Klinik Abteilung fur Elektrophysiologie, Berlin
  - Stadisches Klinikum Brandenburg Med-Klinik I/Kardiologie Pulmologie und Angiologie, Brandenburg
  - Klinikum Coburg II Med. Klinik, Coburg
  - Klinkum Lippe-Detmold Med. Klink II-Kardiologie, Detmold
  - Krankenhaus Duren Medizinische Klinik I Kardiologie/Angiologie, Düren
  - Klinikum Erfurt GmbH, Erfurt
  - Medizinische Universitaetsklinik Innere Medizin III Kardiologie und Angiologie, Frieburg
  - Universitatsklinikum Hamburg-Eppendork Klinik und Poliklinik fur Innere Medizin Abteilung Kardiologie, Hamburg
  - Medizinische Hochschule Innere Medizin/Abt. fur Kardiologie, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Medizinische Universitats-und Ploiklinik Innere Medizin 3, Homburg
  - Klinikum Kassel Medizinische Klinik II, Kassel
  - Universitate zu Koeln Klinik III fur Innere Medizin, Koeln (Lindenthal)
  - Universitat Leipzig Medizinische Klinik und Poliklinik 1 Abteilung fur Kardiologie and Angiolgie, Leipzig
  - Klinikum der Stadt Ludwigshafen Abteilung fur Elektrophysiologie der Kardiologie/Herzzentrum, Ludwigshafen
  - Medizinische Klinik und Poliklnik Innere Medizin C, Mannheim
  - Medizinische Klinik und Poliklinik Innere Medizin C, Münster
  - Klinik am See REHA-Zentrum fur Herz und Kreislauf, Rüdersdorf
  - Medizinische Universitat Tubingen Med. Klinik III, Abt. III fur Kardiologie, Tübingen
  - Reinhard-Nieter-Krankenhaus Med. Klinik 1, Wilhelmshafen
- Hungary (18):
  - State Hospital, Balatonfüred
  - Gottsegen Gyorgy National Institute of Cardiology, Budapest
  - Szent Imre Hospital, Dept. of Internal MedicineI., Budapest
  - Semmelweis University, Dept. of Internal Medicine III., Budapest
  - National Institiute of Pulmonology, Dept. of Cardiology, Budapest
  - Toldi Ferenc Hospital, Dept. of Internal Medicine II., Cegléd
  - Debrecen City Health Service, Debrecen
  - Markoth Ferenc County Hospital, Eger
  - Pandy Kalman Hospital, Gyula
  - County Hospital, Dept. of Internal Medicine I., Kecskemét
  - Miskolc County Hospital, Miskolc
  - Mosonmagyarovar City Karolina Hospital, Mosonmagyaróvár
  - University of Pecs, Cardiology Clinic, Pécs
  - Siofok City Hospital, Siófok
  - Allami Szanatorium, Sopron
  - County Hospital, Dept. of Internal Medicine, Szentes
  - Szent Gyorgy Hospital, Székesfehérvár
  - Markusovszky Hospital, Dept. of Internal Medicine III., Szombathely
- Italy (13):
  - Divisione di Cardiologia Ospedale Civile, Asti
  - Cardiovascular Disease Unit University of Bari-Ploiclinico, Bari
  - Azienda Ospedaliera "Garibaldi S, Luigi Ascoli Tomaselli" Servizio di Cardiologia, Catania
  - Servizio di Cardiologia Azienda Ospedaliera S. Anna, Como
  - Cardiology Division Hospital "Santa Croce e Carle", Cuneo
  - Department of Internal Medicine (DIMI) University of Genova, Genova
  - Ospedale Civile Umberto I Cardiology Division, Mestre
  - S. Paolo Hospital University of Milan Department of Cardiology, Milan
  - Cardiology Unit University of Naples "Frederico II", Napoli
  - Cardiology Unit Policlinico S. Matteo, Pavia
  - Osp. Civile di Piacenza-Div. di Cardiologia, Piacenza
  - Dep. of Cardiovascular and Respiratory Diseases Policlinico Umberto I, Roma
  - Ospedale Umberto I di Torino, Torino
- Netherlands (6):
  - Catharina Ziekenhuis Afd. Cardilolgie, Eindhoven
  - Kennemer Gasthuis, Haarlem
  - Isala Klinieken Locatie De Weezenlanden, JW Zwolle
  - Academisch Ziekenhuis Maastricht Afdeling Cardiologie, Maastricht
  - Department Cardiology Canisius Wilhelmina Hospital, Nijmegen
  - St Elisabeth Ziekenhuis Afdeling Cardiologie, Tilburg
- Poland (20):
  - Klinika Gastroenterologii i Chorob Wewnetrznych Szpital Wojewodzki Zespolony im. Biziela, Ul Ujejskiego 75, Bydgoszcz
  - Oddizial Kardiologii Wojewodzki Szpital Zespolony, Ul Ujejskiego 75, Bydgoszcz
  - Samodzielny Publiczny Szpital Kliniczny Klinika Kardiologii, Bialystok
  - I Klinika Chorob Serca Instytut Kardiologii AM, Gdansk
  - Gornoslaskie Centrum Medyczne I Klinika Kardiologii, Katowice
  - Szpital Wojewodzki Oddzial Kardiologii, Kielce
  - Instytut Kardiologii CMUJ Klinika Choroby Wiencowej, Krakow
  - Oddzial Kardilolgii Wojewodski Szpital Specjalistyczny, Olsztyn
  - Oddzial Kardiologii Wojewodzkie Centrum Medyczne, Opole
  - Oddizial Wewnetzny Szpital Miejski, Ostrowiec Świętokrzyski
  - Oddzial Kardiologii Wojewodzki Szpital Zespolony, Płock
  - Radomski Szpital Specjalistyczny Oddzial Kardiologii, Radom
  - Oddizial Kardiologii Szpital Wojewodzki nr 2, Rzeszów
  - Samodzielny Publiczny Szpital Zespolony Oddizial Kardiologii, Szczecin
  - Wojewodzki Szpital Zespolony Oddzial Kardilolgii, Torun
  - I Klinika Kardiologii CSK WAM, Warsaw
  - Szpital Wolski im. Dr Anny Gostynskiej Oddzial Kardiologii, Warsaw
  - Instytut Kardiologii, Warsaw
  - Klinika Kardiologii IV Wojskowy Szpital Kliniczny, Wroclaw
  - Oddzial Kardiologii Szpital Wojewodzki, Zamość
- Russia (20):
  - Cardiology Department, Moscow Clinical Hospital No. 59, Moscow
  - Res. Inst. of Physical and Chemical Medicine Department of Cardiology Moscow Clinical Hospital No. 29, Moscow
  - Russian State Medical University Clinical facility: Cardiology Department of City Clinical Hospital No. 4, Moscow
  - Moscow State Institute of Peace and Friendship Pharmacology Department, Moscow Clinical Hospital #64, Moscow
  - Cardiology Department Moscow Sechenov Medical Academy, Moscow
  - Medical Centre of General Management Department of the President of the Russian Federation, Cardiology Department Moscow Clinical Hospital No. 51, Moscow
  - Medical Centre of General Management Department of the President of the Russian Federation, Moscow
  - Cardiology Department of State Medical Academy of Postgraduate Education, Myasnikov Clinical Cardiology Research Institute, Moscow
  - Department of Emergency Cardiology Russian Cardiology Research Centre, Moscow
  - Moscow State University of Medicine and Stomatolog, Cardiology Department of Moscow Clinical Hospital No. 50, Moscow
  - Department of Internal Disease No. 5, Moscow State University of Medicine and Stomatology, Cardiology Department Moscow City Hospital No. 11, Moscow
  - Myocardial Infarction Department St Petersburg Hospital, No. 28, Saint Petersburg
  - Cardiology Department, State Research Institute, Saint Petersburg
  - Cardiology Department Alexandrovskiy Hospital, Saint Petersburg
  - Cardiology Department St Petersburg Hospital No. 2, Saint Petersburg
  - Myocardial Infarction Department St Elizabeth Hospital, Saint Petersburg
  - Cardiology Department St. Petersburg State Pavlov Medical University, Saint Petersburg
  - Myocardial Infarction Department St Petersburg Hodpital, No. 29, Saint Petersburg
  - Cardiology Department, St Petersburg Hospital, No. 15, Saint Petersburg
  - Department of Cardiology No. 3 Pokrovskiy Hospital, Saint Petersburg
- Spain (10):
  - Hospital Universitari San Juan Servicio di Cardiologia, Alicante
  - Hospital Valle de Hebron Servicio de Cardiologia, Barcelona
  - Hospital Princeps d'Espanya (Bellvitge) Servicio de cardiologia, Barcelona
  - Hospital Civil De Basurto Cardiology Service, Basurto-Bilbao
  - Hospital Nuestra Senora de Alarcos Unidad de Medicina Intensiva, Ciudad Real
  - Hospital Universitario De Getafe Cardiology Service, Getafe
  - Fundacion Jimenez Diaz Cardiology Service, Madrid
  - Hospital Clinico Universitario San Carlos Servicio de Cardiologia, Madrid
  - Hospital La Paz U.M.Q. de cardiologia, Madrid
  - Hospital de Txagorritxu, Vitoria-Gasteiz